CLINICAL TRIAL: NCT01311544
Title: Evaluation of 4D Magnetic Resonance Angiography (K-t Blast) of Supraortic Vessels in Acute Ischemic Stroke Patients
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2010-A01158-31; LOC/10-11
Record Dates: First submitted 2011-03-07; First posted 2011-03-09 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
The Magnetic Resonance angiography (MRA) of supraaortic vessels is essential for the etiologic of stroke. However, the techniques usually used provide only static evaluation (degree of stenosis, occlusion) but not dynamic. An ultra-fast 3D MRA originally developed for the cardiac imaging, k-t blast (Broad-use Linear Acquisition Speed-up Technique) could be used to review the supraaortic vessels. This MRA offers the following advantages: short acquisition time, wide spatial coverage (of the thoracic aorta to the distal encephalic arteries), 3D spatial resolution and high temporal resolution. These qualities are even more optimal with a high magnetic field (3T). The high temporal resolution is interesting because it provides to repeat a volume every eight seconds and thus to have a dynamic evaluation of vascular filling and to assess the vascular supply of the infarcted territory. This sequence is classified as a 4D MRA.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 years
* Eligibility for intravenous thrombolytic treatment (National Institute of Neurological Disorders and Stroke criteria)
* Permanent ischemic stroke confirm with encephalic MRI (Magnetic Resonance Imaging)
* Patient able of accepting protocol information
* Patient who received information about the protocol and had not expressed its opposition to participate

Exclusion Criteria:

* Pacemaker
* Surgical ferromagnetic clips
* Cochlear implants
* Intraocular metallic foreign body
* Iron implants or objects likely to concentrate the Radio Frequency field
* Claustrophobia
* Known intolerance to contrast media (DOTAREM)
* Pregnant women (Beta Human Chorionic gonadotrophin performed for biological assessment of thrombolysis)
* Patient with severe kidney with Glomerular Filtration rate < 30 ml/min
* Persons subject to major legal protection (safeguarding justice, guardianship, trusteeship), persons deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute ischemic stroke
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2011-03

PRIMARY OUTCOMES:
Images quality for each cervical and intracranial arteries | 6 months

SECONDARY OUTCOMES:
Quantification of carotid stenosis with NASCET classification | 6 months
Study of dynamic vascular consequences of carotid stenosis | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: jean-yves gauvrit, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, Brittany Region, France